CLINICAL TRIAL: NCT00400439
Title: A Phase II, Placebo-Controlled, Double-Blind Extension Study of Study NC19453 Assessing Long-term Safety and Efficacy of RO4607381
Brief Title: A Long Term Extension of Study NC19453 Evaluating Safety and Efficacy of RO4607381
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NC20716
Record Dates: First submitted 2006-11-15; First posted 2006-11-16 (Estimated); Results first posted 2020-01-03 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease | interventions — dalcetrapib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- dalcetrapib (RO4607381) (Experimental)
  Interventions: Drug: dalcetrapib (RO4607381)
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: dalcetrapib (RO4607381) — 900mg po daily for 24 weeks
  Arms: dalcetrapib (RO4607381)
Drug: placebo — po daily for 24 weeks
  Arms: placebo

SUMMARY:
This 2 arm study will assess the long term safety and efficacy of RO4607381 in patients with coronary heart disease or a coronary heart disease (CHD) risk equivalent who have completed study NC19453. Patients eligible to participate in the extension study will continue on the treatment they were originally assigned to ie RO4607381 (900mg po) or placebo daily, with concomitant daily atorvastatin (10 to 80mg po). The anticipated time on study treatment is 6 months post study NC19453, and the target sample size is approximately 100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* patients who have completed treatment on study NC19453.

Exclusion Criteria:

* any significant lymph node abnormalities at the end of study NC19453.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- United States (8):
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Louisville, Kentucky
  - Bethesda, Maryland
  - Minneapolis, Minnesota
  - Statesville, North Carolina
  - Cincinnati, Ohio
  - Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dalcetrapib (RO4607381) | Placebo
Started | 52 | 25
Completed | 47 | 23
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dalcetrapib (RO4607381) | Placebo | Total
Number analyzed (Participants) | 52 | 25 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (7.03) | 60.8 (7.83) | 60.6 (7.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 3 | 15
  Male | 40 | 22 | 62

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in HDL-C
Time Frame: Baseline and Week 24 (Week 48 from start of NC19453(NCT00353522))
Measure: Least Squares Mean (Standard Error); unit: Percentage Change of HDL-C
Arm/Group | Dalcetrapib (RO4607381) | Placebo
Number analyzed (Participants) | 52 | 25
Percentage Change of HDL-C | 33.76 (4.43) | 3.69 (5.81)

2. Secondary Outcome: Change From Baseline in High Density Lipoprotein Cholesterol (HDL-C), Total Cholesterol (TC), Low Density Lipoprotein Cholesterol (LDL-C), Triglycerides (TG), Apolipoprotein B (ApoB) and Apolipoprotein A1 (ApoA1)
Time Frame: Baseline and Week 24 (Week 48 from start of NC19453)
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Dalcetrapib (RO4607381) | Placebo
Number analyzed (Participants) | 52 | 25
mg/dL
  HDL-C | 37.29 (5.11) | 2.98 (6.08)
  Total Cholesterol | 16.60 (5.17) | -0.96 (6.16)
  LDL-C | 7.54 (5.12) | 2.16 (6.13)
  Triglycerides | 2.95 (21.44) | -8.10 (25.91)
  ApoB | 4.02 (3.36) | -0.79 (4.09)
  ApoA1 | 25.13 (3.55) | 8.91 (4.28)

ADVERSE EVENTS:
Description: Study was an extension of NC19453. Adverse Event data was not collected.
Arm/Group | Dalcetrapib (RO4607381) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No